CLINICAL TRIAL: NCT02973048
Title: Hyperbaric Bupivacaine Versus Hyperbaric Prilocaine 2% for Cesarean Section Under Spinal Anesthesia: a Randomised Clinical Trial
Brief Title: Hyperbaric Bupivacaine Versus Hyperbaric Prilocaine 2% for Cesarean Section Under Spinal Anesthesia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Saint Pierre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: B076201627677
Record Dates: First submitted 2016-07-25; First posted 2016-11-25 (Estimated); Results first posted 2020-07-02 (Actual); Last update posted 2020-07-02 (Actual); Status verified 2020-07

CONDITIONS: Pregnant Women; Pain; Hypotension
Keywords: Cesarean delivery; Spinal anesthesia; Local anesthetics
MeSH Terms: conditions — Pain; Hypotension | interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hyperbaric bupivacaine (Placebo Comparator): Hyperbaric bupivacaine 0.5% will be administered at the dose of 10 mg intrathecally associated with 100 µg of morphine and 2.5 µg of sufentanyl.
  Interventions: Drug: Hyperbaric bupivacaine
- Hyperbaric prilocaine (Active Comparator): Hyperbaric prilocaine 2% will be administered at the dose of 50 mg intrathecally associated with 100 µg of morphine and 2.5 µg of sufentanyl.
  Interventions: Drug: Hyperbaric prilocaine

INTERVENTIONS:
Drug: Hyperbaric bupivacaine — The dose of 10 mg of hyperbaric bupivacaine will be administered to one of two groups intrathecally and the quality of sensory and motor block as well as side-effects will be observed at precise time points.
  Other Names: Marcaine
  Arms: Hyperbaric bupivacaine
Drug: Hyperbaric prilocaine — The dose of 50 mg of hyperbaric prilocaine will be administered to one of two groups intrathecally and the quality of sensory and motor block as well as side-effects will be observed at precise time points.
  Other Names: Tachipri
  Arms: Hyperbaric prilocaine

SUMMARY:
Over the past 15 years, cesarean delivery is most commonly performed under spinal anesthesia using hyperbaric bupivacaine which provides an adequate sensory and motor block. Despite effective surgical anesthesia, bupivacaine is associated with long duration motor block and dose-dependent maternal hypotension potentially harmful for the fetus. Prilocaine with its new 2% hyperbaric formulation (HP), developed recently, showed rapid onset of action and faster regression of motor block compared to other local anesthetics without noteworthy side-effects when used intrathecally. The aim of this randomized, multicenter, powered clinical trial is to investigate whether HP may be an efficient alternative to hyperbaric bupivacaine for scheduled caesarean delivery under spinal anesthesia, with more rapid rehabilitation and less adverse effects. Our hypothesis is that hyperbaric prilocaine offers shorter motor block and more rapid rehabilitation than bupivacaine.

ELIGIBILITY:
Inclusion Criteria :

* American Society of Anesthesiologists physical status (ASA) < III
* Age 18-40 year
* Body Weight <110 kg
* Height between 160 and 175 cm
* Gestational age>37 SA
* Elective cesarean delivery
* Singleton pregnancy
* Non complicated pregnancy
* Signed informed consent obtained prior to any study specific assessments and procedures

Exclusion Criteria:

* Twin pregnancy
* History of 2 cesarean section or more
* Diabetes and gestational diabetes
* Placenta praevia
* Congenital foetal abnormality
* Intrauterine growth retardation
* Patient in labour
* Membrane rupture
* Known allergy to local anaesthetics
* Standard contraindications to neuraxial block.
* Disagreement of the patient
* Neurological impairment
* Gestational low blood pressure
* Pre eclampsia and eclampsia

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2018-03-12 (Actual); Primary Completion 2018-11-08 (Actual); Study Completion 2018-11-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Panayota KAPESSIDOU, MD, PhD, Study Director — University Hospital Saint-Pierre (CHU Saint-Pierre), Université Libre de Bruxelles (ULB); Philippe GOFFARD, MD, Principal Investigator — University Hospital Saint-Pierre (CHU Saint-Pierre), Université Libre de Bruxelles (ULB)
Locations (2):
- Belgium (2):
  - University Hospital Saint-Pierre, Université Libre de Bruxelles (ULB), Brussels, Brussels Capital
  - Clinique Ste-Anne/St-Remi, Anderlecht

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gautier P, De Kock M, Huberty L, Demir T, Izydorczic M, Vanderick B. Comparison of the effects of intrathecal ropivacaine, levobupivacaine, and bupivacaine for Caesarean section. Br J Anaesth. 2003 Nov;91(5):684-9. doi: 10.1093/bja/aeg251. PMID 14570791
- [Background] Guntz E, Latrech B, Tsiberidis C, Gouwy J, Kapessidou Y. ED50 and ED90 of intrathecal hyperbaric 2% prilocaine in ambulatory knee arthroscopy. Can J Anaesth. 2014 Sep;61(9):801-7. doi: 10.1007/s12630-014-0189-7. Epub 2014 Jun 7. PMID 24906303
- [Background] Guntz E, Kapessidou Y. Spinal prilocaine for same-day surgery: the importance of equipotent doses. Can J Anaesth. 2016 Aug;63(8):985-6. doi: 10.1007/s12630-016-0645-7. Epub 2016 Apr 4. No abstract available. PMID 27044397
- [Derived] Goffard P, Leloup R, Vercruysse Y, Fils JF, Gautier PE, Kapessidou Y. Comparison of equipotent doses of intrathecal hyperbaric prilocaine 2% and hyperbaric bupivacaine 0.5% for elective caesarean section: A prospective, randomised, controlled, two-centre clinical trial. Eur J Anaesthesiol. 2022 Mar 1;39(3):227-235. doi: 10.1097/EJA.0000000000001548. PMID 34101713

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All participants were recruited at CHU Saint-Pierre and Sainte-Anne Saint-Rémy hospitals (Brussels). Of 88 patients assessed for eligibility, only 40 were randomized to treatment (17 not meeting inclusion criteria and 31 declined to participate)
Period: Overall Study
Arm/Group | Hyperbaric Bupivacaine | Hyperbaric Prilocaine
Started | 20 | 20
Completed | 19 | 17
Not Completed | 1 | 3
Not completed — Epidural catheter insertion failure | 1 | 0
Not completed — Withdrawal by Subject | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Hyperbaric Bupivacaine | Hyperbaric Prilocaine | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 36.5 [32 to 38] | 32 [28.75 to 35.25] | 36 [29.75 to 38]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 20 | 40
  Male | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Weight [Mean (Standard Deviation); unit: kg] | 74.8 (12.85) | 76.2 (13.4) | 75.5 (12.98)
Height [Median (Inter-Quartile Range); unit: cm] | 164 [161 to 166.25] | 164 [160 to 168.25] | 164 [160 to 167.25]
BMI [Median (Inter-Quartile Range); unit: kg/m^2] | 26.37 [23.77 to 30.58] | 26.19 [24.75 to 30.58] | 26.26 [24.61 to 30.58]
American Society of Anesthesiologists physical status (ASA) II [Count of Participants; unit: Participants] — The American Society of Anesthesiologists (ASA) physical status classification system was developed to offer clinicians a simple categorization of a patient's physiological status that can be helpful in predicting operative risk.
  ASA 1: Normal healthy patient, ASA 2: Patient with a mild systemic disease ASA 3: Patient with a severe systemic disease not life-threatening ASA 4: Patient with a severe systemic disease being a constant threat to life. ASA 5: Moribund patient
  Pregnancy of > 20 amenorrhea age is considered an ASA II grade; parturients of ASA > II were excluded from study
  Participants | 20 | 20 | 40
Gestational Age (GA) [Median (Inter-Quartile Range); unit: weeks] | 39 [38 to 39] | 39 [38 to 39] | 39 [38 to 39]
Gestity [Median (Inter-Quartile Range); unit: Pregnancies] | 2 [2 to 3] | 2 [2 to 3] | 2 [2 to 3]
Parity [Median (Inter-Quartile Range); unit: Deliveries] | 1 [0 to 1] | 1 [0 to 1] | 1 [0 to 1]
Previous c-Section [Number; unit: Participants] | 13 | 6 | 19

OUTCOME MEASURES:

1. Primary Outcome: Time to Regression of Motor Block
Description: Time to regression of motor block is the time between maximal blockade (score 1, as evaluated by the Modified Bromage scale), and no blockade (score 6). Degree of motor blockade is assessed before and 10, 15, 20 minutes after spinal anesthesia, then every 15 minutes until the end of surgery, and thereafter, every 30 minutes until complete regression of motor block
Time Frame: until complete regression of motor block (up to 4 hours)
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | Hyperbaric Bupivacaine | Hyperbaric Prilocaine
Number analyzed (Participants) | 19 | 17
minutes | 180 [142.5 to 239.5] | 130 [120 to 166]

2. Secondary Outcome: Time to Successful Anesthesia (Successful Sensory Block)
Description: Time between spinal injection and reached bilateral T4 sensory level.
Time Frame: From spinal injection of the local anesthetic to bilateral T4 level (average 20 minutes)
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Hyperbaric Bupivacaine | Hyperbaric Prilocaine
Number analyzed (Participants) | 19 | 17
minutes | 9.63 (3.48) | 11.18 (2.7)

3. Secondary Outcome: Number of Participants Per Maximal Level of Sensory Block Attained After Spinal Anesthesia
Description: Level of Sensory block is assessed as loss of sensation to cold, and represents the dermatomal level under which anesthesia is effective. It is measured every 2 minutes after spinal anesthesia during 15 minutes, then every 5 minutes until the end of surgery, thereafter, once 30 minutes until total regression of sensory block (T12-S1). A dermatome is the area of skin that is supplied by a single spinal nerve - Dermatome levels : C5-C8 for Cervical levels and T1-T4 for Thoracic levels.
  To perform cesarean section loss of cold sensation at a dermatome of at least T4 has to be obtained.
  The results are expressed as the number of patients reaching each dermatomal level from T4 and above (see below) as maximal sensory level, this is a usual outcome used to evaluate the quality of anesthesia.
Time Frame: until complete release of sensory block (T12-S1) (average 4 hours)
Measure: Count of Participants; unit: Participants
Arm/Group | Hyperbaric Bupivacaine | Hyperbaric Prilocaine
Number analyzed (Participants) | 19 | 17
Participants
  Sensory level dermatome C5 | 0 | 1
  Sensory level dermatome C6 | 3 | 1
  Sensory level dermatome C7 | 0 | 0
  Sensory level dermatome C8 | 2 | 1
  Sensory level dermatome T1 | 0 | 0
  Sensory level dermatome T2 | 4 | 2
  Sensory level dermatome T3 | 7 | 6
  Sensory level dermatome T4 | 3 | 6

4. Secondary Outcome: Time to Resolution of Sensory Block
Description: Evaluation at every 2 minutes after spinal anesthesia during 15 minutes, then every 5 minutes until the end of surgery, and thereafter, every 30 minutes until total regression of sensory block (T12-S1).
Time Frame: until complete release of sensory block (T12-S1) (average 4 hours)
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Hyperbaric Bupivacaine | Hyperbaric Prilocaine
Number analyzed (Participants) | 19 | 17
minutes | 212.95 (51.48) | 169.59 (32.71)

5. Secondary Outcome: Time to Motor Block Onset
Description: Time of installation of the motor block (time between spinal injection and maximum motor block of 1, as evaluated by the Modified Bromage scale). Degree of motor blockade is assessed before and 10, 15, 20 minutes after spinal anesthesia
Time Frame: From spinal injection of the local anesthetic to bilateral T4 level and during surgery (average 1 hour)
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | Hyperbaric Bupivacaine | Hyperbaric Prilocaine
Number analyzed (Participants) | 19 | 17
minutes | 16 [10 to 16] | 10 [10 to 16]

6. Secondary Outcome: Number of Patients With Hypotension and Use of Vasopressors
Description: Arterial blood pressure will be measured at every 1 minute during the first 15 minutes, then at every 2.5 minutes until the end of surgery, and at every 20 minutes in the Post Anesthesia Care Unit (PACU). A low blood pressure (hypotension) is defined as a systolic blood pressure lower than 20% or more than the basal blood pressure (Systolic blood pressure before spinal anesthesia)
Time Frame: up to 2 hours after surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Hyperbaric Bupivacaine | Hyperbaric Prilocaine
Number analyzed (Participants) | 19 | 17
Participants
  Hypotension | 17 | 9
  Vasopressors use | 16 | 10

7. Secondary Outcome: Number of Participants With Urinary Retention
Description: All parturients will be questioned and examined for urinary retention (yes or no)
Time Frame: up to 4 hours after surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Hyperbaric Bupivacaine | Hyperbaric Prilocaine
Number analyzed (Participants) | 19 | 17
Participants | 2 | 2

8. Secondary Outcome: Time to First Walk
Description: Time for the patients to be able to walk in their room then in the hallway without any assistance for the first time.
Time Frame: up to 24h after surgery
Measure: Median (Inter-Quartile Range); unit: Minutes
Arm/Group | Hyperbaric Bupivacaine | Hyperbaric Prilocaine
Number analyzed (Participants) | 19 | 17
Minutes | 318 [194 to 420] | 198 [175.5 to 250.75]

9. Secondary Outcome: Maternal Satisfaction Assessed by Visual Analogic Scale (VASS)
Description: All patients will be asked to rate their satisfaction about anesthetic technique during surgery and in the arrival in the Post Anesthesia Care Unit (PACU). Satisfaction evaluated by Visual analog scale (0 cm= very unsatisfied and 10cm = very satisfied)
Time Frame: up to 24 hours after surgery
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Hyperbaric Bupivacaine | Hyperbaric Prilocaine
Number analyzed (Participants) | 19 | 17
score on a scale | 9 [8 to 9] | 9 [8 to 9.25]

10. Secondary Outcome: Maternal Rehabilitation Assessed by Visual Analogic Scale (VASR)
Description: Maternal rehabilitation is evaluated at postoperative Day1, postoperative Day 2 and postoperative Day 3. Evaluation by Visual analog scale (0 cm= very poor and 10cm = excellent)
Time Frame: up to 72 hours after surgery
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Hyperbaric Bupivacaine | Hyperbaric Prilocaine
Number analyzed (Participants) | 19 | 17
score on a scale | 9 [7 to 10] | 9 [8 to 9.25]

11. Secondary Outcome: Number of Participants With Adverse Events (Nausea, Vomiting, Pruritis, Headache)
Description: Evaluation from 15 minutes after spinal injection to the end of surgery, then every 4 hours for 24 hours, then once a day for 3 days (score 0=no symptom; 1=symptom with no necessary treatment; 2=symptom present and treated)
Time Frame: up to 72 hours after surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Hyperbaric Bupivacaine | Hyperbaric Prilocaine
Number analyzed (Participants) | 19 | 17
Participants
  Peroperative: score 0 (no symptom) | 18 | 13
  Peroperative: score 1 (symptom with no necessary treatment) | 1 | 1
  Peroperative: score 2 (symptom present and treated) | 0 | 3
  Day 0: score 0 (no symptom) | 14 | 12
  Day 0: score 1 (symptom with no necessary treatment) | 4 | 5
  Day 0: score 2 (symptom present and treated) | 1 | 0
  Day 1: score 0 (no symptom) | 16 | 17
  Day 1: score 1 (symptom with no necessary treatment) | 3 | 0
  Day 1: score 2 (symptom present and treated) | 0 | 0
  Day 2: score 0 (no symptom) | 18 | 17
  Day 2: score 1 (symptom with no necessary treatment) | 1 | 0
  Day 2: score 2 (symptom present and treated) | 0 | 0
  Day 3: score 0 (no symptom) | 18 | 17
  Day 3: score 1 (symptom with no necessary treatment) | 1 | 0
  Day 3: score 2 (symptom present and treated) | 0 | 0

12. Secondary Outcome: Number of Participants With Transient Neurologic Symptoms (TNS)
Description: Evaluation of apparition of TNS at postoperative Day 1, postoperative Day 2, postoperative Day 3 and postoperative Day 15. TNS are defined as pain and/or dysesthesia occurred after complete release of sensory block at the gluteal level, at the thighs and at the legs.
Time Frame: up to 15 Days after surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Hyperbaric Bupivacaine | Hyperbaric Prilocaine
Number analyzed (Participants) | 19 | 17
Participants | 0 | 0

13. Secondary Outcome: Pain as Assessed by Visual Analogue Scale
Description: Pain levels will be determined at incision, baby delivery, peritoneal and skin closure, every 5 minutes during surgery, and thereafter every 4 hours for 24 hours. Visual analog pain score (scale = 0 no pain; 10 = worst pain imaginable). Patient will receive additional analgesic treatment above VAS>3.
Time Frame: up to 24 hours after surgery
Population: VAS are presented only at 1 Hour, 2 Hours , 3 Hours and 4 Hours post-surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Hyperbaric Bupivacaine | Hyperbaric Prilocaine
Number analyzed (Participants) | 19 | 17
Participants
  VAS at 1 Hour: VAS=0 (no pain) | 13 | 7
  VAS at 1 Hour: VAS 1-2 (No additional analgesic treatment) | 6 | 9
  VAS at 1 Hour: VAS >3 (additional analgesic treatment) | 0 | 1
  VAS at 2 Hours: VAS=0 (no pain) | 11 | 3
  VAS at 2 Hours: VAS 1-2 (No additional analgesic treatment) | 6 | 13
  VAS at 2 Hours: VAS >3 (additional analgesic treatment) | 2 | 1
  VAS at 3 Hours: VAS=0 (no pain) | 9 | 9
  VAS at 3 Hours: VAS 1-2 (No additional analgesic treatment) | 7 | 6
  VAS at 3 Hours: VAS >3 (additional analgesic treatment) | 3 | 2
  VAS at 4 Hours: VAS=0 (no pain) | 10 | 12
  VAS at 4 Hours: VAS 1-2 (No additional analgesic treatment) | 7 | 5
  VAS at 4 Hours: VAS >3 (additional analgesic treatment) | 2 | 0

14. Secondary Outcome: Newborn Apgar Score
Description: Newborn Apgar score assessed at 1, 5, 10 minutes after baby extraction. The Apgar score is determined by evaluating the newborn baby on five simple criteria on a scale from 0 to 2, then summing up the five values thus obtained. The overall resulting score ranges from 0 to 10 ( 0-3 : severely depressed, 4-6 : Moderately depressed and 7-10 : Excellent condition).
  The five criteria are summarized using words chosen to form an abbreviation (Appearance, Pulse, Grimace, Activity, Respiration).
Time Frame: up to 10 minutes after baby extraction
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Hyperbaric Bupivacaine | Hyperbaric Prilocaine
Number analyzed (Participants) | 19 | 17
score on a scale
  Apgar at 1 minute | 9 [9 to 9] | 9 [9 to 9]
  Apgar at 3 minutes | 10 [10 to 10] | 10 [10 to 10]
  Apgar at 5 minutes | 10 [10 to 10] | 10 [10 to 10]

15. Secondary Outcome: Newborn Methemoglobinemia (MetHb)
Description: Newborn Methemoglobinemia (MetHb) will be assessed at delivery by cordal blood sample, as a routine control in obstetrics, and expressed as a percentage of total hemoglobinemia.
  Methemoglobinemia (MetHb) is a blood disorder in which an abnormal amount of methemoglobin (hemoglobin in the form metalloprotein) is produced. This specific type of of Hemoglobin carries oxygen through your blood but doesn't release it to the cells.
Time Frame: average 1 hour
Measure: Median (Inter-Quartile Range); unit: percentage of MetHb
Arm/Group | Hyperbaric Bupivacaine | Hyperbaric Prilocaine
Number analyzed (Participants) | 19 | 17
percentage of MetHb | 1.8 [1.7 to 1.9] | 1.7 [1.6 to 1.9]

16. Secondary Outcome: Newborn Umbilical pH
Description: Newborn umbilical pH will be assessed at delivery by cordal blood sample, as a routine control, and expressed as standard value
Time Frame: average 1 hour
Measure: Median (Inter-Quartile Range); unit: pH
Arm/Group | Hyperbaric Bupivacaine | Hyperbaric Prilocaine
Number analyzed (Participants) | 19 | 17
pH | 7.33 [7.29 to 7.34] | 7.32 [7.29 to 7.33]

17. Secondary Outcome: Time of Surgery
Description: Time between incision and end of surgery
Time Frame: average 1 hour
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | Hyperbaric Bupivacaine | Hyperbaric Prilocaine
Number analyzed (Participants) | 19 | 17
minutes | 45 [40.5 to 56.5] | 50 [44 to 54]

18. Secondary Outcome: Time From Spinal Injection to Baby Delivery
Description: Time between spinal injection and baby delivery
Time Frame: average 1 hour
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | Hyperbaric Bupivacaine | Hyperbaric Prilocaine
Number analyzed (Participants) | 19 | 17
minutes | 24 [22 to 27] | 25 [24 to 27]

19. Secondary Outcome: Time From Baby Delivery to End of Surgery
Description: Time between baby delivery, and the end of surgery
Time Frame: average 1 hour
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Hyperbaric Bupivacaine | Hyperbaric Prilocaine
Number analyzed (Participants) | 19 | 17
minutes | 36.68 (10.19) | 38.24 (6.55)

20. Secondary Outcome: Total Blood Loss
Description: Total blood loss (milliliters) during surgery
Time Frame: average 1 hour
Measure: Median (Inter-Quartile Range); unit: milliliters
Arm/Group | Hyperbaric Bupivacaine | Hyperbaric Prilocaine
Number analyzed (Participants) | 19 | 17
milliliters | 415 [312.5 to 746.25] | 485 [305 to 562.5]

21. Secondary Outcome: Obstetrician Satisfaction
Description: Satisfaction ranged between 1 (totally unsatisfied) to 4 (totally satisfied) assessed at the end of surgery
Time Frame: average 1 hour
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Hyperbaric Bupivacaine | Hyperbaric Prilocaine
Number analyzed (Participants) | 19 | 17
score on a scale | 4 [4 to 4] | 4 [4 to 4]

22. Secondary Outcome: Midwife Satisfaction
Description: Satisfaction ranged between 1 (totally unsatisfied) to 4 (totally satisfied) assessed at postoperative Day 3
Time Frame: 72 hours after surgery
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Hyperbaric Bupivacaine | Hyperbaric Prilocaine
Number analyzed (Participants) | 19 | 17
score on a scale | 3 [1.5 to 4] | 4 [3 to 4]

ADVERSE EVENTS:
Time Frame: Adverse event were collected from spinal injection until 15 Days following the day of surgery.
Arm/Group | Hyperbaric Bupivacaine | Hyperbaric Prilocaine
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/17
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/17
Other Adverse Events (participants affected / at risk) | 8/19 | 8/17
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Hyperbaric Bupivacaine (N=19) | Hyperbaric Prilocaine (N=17)
Transient neurologic symptoms (Nervous system disorders) | 1 | 1
Nausea (Gastrointestinal disorders) | 8 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-11-02): https://cdn.clinicaltrials.gov/large-docs/48/NCT02973048/Prot_SAP_000.pdf